CLINICAL TRIAL: NCT06026579
Title: Clinical Characteristics and Subgroups in Greater Trochanteric Pain Syndrome
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: NHS Research Scotland (Other)
Responsible Party: Sponsor
Other Study IDs: GN23PY207
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Greater Trochanteric Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This cross-sectional study will gather participant data from clinical assessment and questionnaires for individuals with a clinical diagnosis of Greater Trochanteric Pain Syndrome.

DETAILED DESCRIPTION:
Greater trochanteric pain syndrome (GTPS) is characterised by pain over and around the greater trochanter and is primarily due to gluteal tendinopathy. Pain associated with GTPS can affect an individual's ability to perform daily activities while also having a negative impact on sleep, work and participation in sport. Quality of life is often impaired and comparable to severe hip osteoarthritis. A significant number report chronic pain and disability with 29% and 45% of individuals continuing to experience pain at five and 11-year follow-up respectively.

Exercise programmes which specifically target the gluteal muscles and tendons are normally the first-line treatment for GTPS, however 20-50% of individuals do not fully recover within 12 months with this intervention. The reasons for this poor response remain unclear but may be associated with the presence of certain clinical characteristics. Diabetes, obesity, co-existing musculoskeletal disorders, psychological factors and physical activity level may affect prognosis and treatment outcome in GTPS. Co-existing low back and/or hip joint pain is common in this population and a higher number of pain sites has been associated with poorer outcome in other musculoskeletal conditions. In clinical trials, participants with GTPS are often grouped together regardless of individual clinical characteristics. Current treatment strategies appear inadequate for a proportion of patients with this condition meaning alternative options are required to achieve a positive clinical outcome.

Subgroups of patients within the same condition have been identified in low back pain, osteoarthritis and patellofemoral pain. Thus, it is important to look for subgroups within the clinically diagnosed GTPS population.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged > 18 years who currently reside within Greater Glasgow and Clyde
* Lateral hip pain of any duration
* Able to give written informed consent
* Pain on direct palpation of the gluteal tendon insertion on the greater trochanter and additionally at least one of the following pain provocation tests must also be positive:

  1. FABER (Flexion, Abduction, External Rotation of the hip)
  2. FADER (Flexion, Adduction, External Rotation of the hip)
  3. FADER and resisted Internal Rotation (IR) (FADER position plus resisted IR of the hip)
  4. Single leg stand for 30 seconds
  5. Resisted hip abduction at end-range adduction

Exclusion Criteria:

* Lateral hip pain secondary to another source e.g. hip joint pathology or lumbar referred pain
* Inflammatory joint conditions
* Neurological conditions
* Pregnancy
* Unable or unwilling to give informed consent
* Unable to write, read or comprehend English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a clinical diagnosis of GTPS will be recruited from NHS physiotherapy waiting lists in Greater Glasgow and Clyde and also from the general public who currently reside in Greater Glasgow and Clyde.
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline and 12 months
  The NPRS is a unidimensional measure of pain intensity.Worst and average lateral hip pain over past week will be measured on an 11-point scale between 0 (no pain) and 10 (worst pain imaginable).
Patient Specific Functional Scale (PSFS) | Baseline and 12 months
  Function will be assessed using the PSFS. Each participant will identify three activities they are unable to perform or have difficulty performing due to their problem. They rate the difficulty on a scale from 0 (unable to perform) to 10 (able to perform at prior level). I
Victoria Institute of Sports Assessment-GTPS (VISA-G) | Baseline and 12 months
  Disability will be measured using the VISA-G questionnaire It is currently the preferred option to capture the disability associated with GTPS and has previously been validated for use in this condition.
Tampa Scale for Kinesiophobia (TSK-17) | Baseline and 12 months
  The TSK-17 is a 17-item questionnaire used to assess fear of movement and reinjury. Four-point Likert scales are used. Total scores range from 17 to 68 with a score greater than 37 indicating kinesiophobia.
Depression and Anxiety Stress Scales-21 (DASS-21) | Baseline and 12 months
  Anxiety and depression will be measured using the DASS-21 questionnaire.The DASS items are scored on a 4-point scale ranging from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). Higher scores indicate more frequent symptomatology.
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline and 12 months
  PSEQ is a 10-item questionnaire which measures a person's beliefs about whether they can engage in activities and enjoy life despite experiencing pain. Participants rate how confidently they can perform each activity on a 7-point Likert scale. The total score ranges from 0 to 60, where higher scores reflect stronger self-efficacy.
Euro Qol (EQ-5D-5L) | Baseline and 12 months
  The EQ-5D-5L is a five-dimension questionnaire for measuring health-related quality of life. Participants rate their health status on five dimension; mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of these five dimensions has five statements and each participant will tick one of five boxes for each dimension. An index value (0-1) is calculated from five separate questions. A score of 1 reflects greater quality of life. Each participant also evaluates their current overall health status using a visual analogue scale with a score of 0 indicating the worst imaginable health and a score of 100 the best imaginable health.
International Physical Activity Questionnaire - Short Form (IPAQ-SF) | Baseline and 12 months
  The IPAQ-SF is a widely used questionnaire to measure physical activity. The seven questions relate to the amount of time the participant has spent being physically active in the previous 7 days. It covers the domains of leisure time, work-related, transport related and domestic and gardening activities.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Clifford, PhD, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No